CLINICAL TRIAL: NCT03748771
Title: Validation of ApneaLink Air Home Sleep Testing in the Diagnosis of Obstructive Sleep Apnea in Adolescent Children
Status: Completed | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCSD 171173
Record Dates: First submitted 2018-11-12; First posted 2018-11-21 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- ApneaLink Air (Experimental): Half of the participants will undergo HST no greater than one week prior to their in-laboratory PSG, while the other half will undergo HST no greater than one week following their in laboratory PSG. All participants will also undergo their HST concurrent to their in-laboratory PSG. The rational for splitting participants in these two groups is to equally distribute the effects of the first night evenly, in which the sleep architecture including reduced total rapid eye movement (REM) sleep time can vary during the first ever sleep study. As the HST will be compared to the in-lab PSG, we would like to evenly distribute this effect by having two groups of ten participants.
  Interventions: Device: ApneaLink Air

INTERVENTIONS:
Device: ApneaLink Air — The ApneaLink Air device is indicated for use by Health Care Professionals (HCP), where it may aid in the diagnosis of sleep disordered breathing for adult patients.
  ApneaLink Air records the following data: patient respiratory nasal airflow, snoring, blood oxygen saturation, pulse and respiratory effort during sleep. The device uses these recordings to produce a report for the HCP that may aid in the diagnosis of sleep disordered breathing or for further clinical investigation. The device is intended for home and hospital use under the direction of a HCP.

SUMMARY:
The feasibility and the validity of the ApneaLink Air home sleep testing (HST) device will be tested in adolescent children. The ApneaLink Air HST device is cleared for the diagnosis of obstructive sleep apnea (OSA) in adults..

DETAILED DESCRIPTION:
Obstructive sleep apnea is highly prevalent in children affecting 2-3% of children and up to 10% of obese children. The reported prevalence is likely underestimated due to the lack of available laboratory polysomnography (PSG) testing for children. The high prevalence of OSA coupled with an increase in obesity, a major risk factor of OSA in children, has resulted in a significant strain for in laboratory PSG including children in the greater San Diego county. Currently, HST in children is restricted based on the limited availability of HST devices on children that have attained clearance by the US Food and Drug Administration (FDA). In this study, the feasibility and the validity of the ApneaLink Air HST device will be tested in children 12 years old and over. The ApneaLink Air HST device is cleared for the diagnosis of OSA in adults and is frequently used amongst adult sleep medicine physicians. Adolescent children will be recruited whose clinically indicated in laboratory PSG will be performed at Rady Children's Hospital. Concurrent to their in-laboratory PSG, they will have their sleep assessed using the ApneaLink Air device. Ten children will repeat the ApneaLink Air HST at home following their sleep study within one week, and the remaining ten children will have their ApneaLink Air HST performed within one week prior to their in laboratory clinically indicated PSG.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptoms of OSA needing a sleep study
* Patients between the ages of 12 and 17 years, inclusive

Exclusion Criteria:

* Patients less than 12 years old
* Patients 18 years old or older
* Children with syndromes or congenital disease including Down Syndrome, Prader-Willi syndrome, children with craniofacial disorders, and finally children with congenital heart disease or pulmonary hypertension

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhattacharjee R, Benjafield A, Blase A, Dever G, Celso J, Nation J, Good R, Malhotra A. The accuracy of a portable sleep monitor to diagnose obstructive sleep apnea in adolescent patients. J Clin Sleep Med. 2021 Jul 1;17(7):1379-1387. doi: 10.5664/jcsm.9202. PMID 33666166

RESULTS

PARTICIPANT FLOW:
Groups:
- ApneaLink Air Cohort: Patients underwent HST no greater than one week prior to or following their in-lab PSG.
Period: Overall Study
Arm/Group | ApneaLink Air Cohort
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ApneaLink Air Cohort: Patients underwent HST (home sleep apnea testing) no greater than one week prior to or following their in-lab PSG.
Arm/Group | ApneaLink Air Cohort
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 7
  Hispanic | 11
  Pacific Islander | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
BMI [Mean (Standard Deviation); unit: kg/square meters] | 32 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of HST Compared to ALT (ApneaLink Lab Testing) and PSG (Polysomnography)
Description: Accuracy is measured by ODI (oxygen desaturation index) and AHI (apnea hypopnea index)
  The ODI is defined as the number of episodes of oxygen desaturation per hour of sleep, with oxygen desaturation defined as a decrease in blood oxygen saturation (SpO2) to lower than 3% below baseline. The ODI is presented as an index to indicate the number of oxygen dips per hour of sleep.
  The AHI indicates the number of apneas or hypopneas which occured during the sleep study, divided by the hours of sleep. The AHI is an Index which indicates how many events occurred each hour
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | ApneaLink Air Cohort
Number analyzed (Participants) | 20
events per hour
  AHI from HST | 6.2 (10.7)
  ODI from HST | 10.9 (11.4)
  AHI from ALT | 11.6 (21.8)
  ODI from ALT | 16.9 (24.0)
  AHI from PSG | 18.6 (35.8)
  ODI from PSG | 13.5 (26.7)

2. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with the HST and PSG procedures were determined by interview. Question read: "Do you prefer HST over PSG?"
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | ApneaLink Air Cohort
Number analyzed (Participants) | 17
Participants
  Yes | 12
  No | 4
  No Difference | 1

3. Secondary Outcome: Number of Successful HST Evaluations
Description: An unsuccesful HST or HST failure will be defined as:
  1. Loss of the nasal flow channel, or thoracic or abdominal sensor
  2. Recordings with less than 4h of artifact-free recording time
  3. Less than 4h of Sp02 signal
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | ApneaLink Air Cohort
Number analyzed (Participants) | 20
Participants
  Successful HST | 15
  Successful ALT | 17

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study. For each patient this began from when they were enrolled in the study, and was completed when they finished all study activities including the home sleep test. The duration of each patients enrollment in the study was <7 days.
Arm/Group | ApneaLink Air Cohort
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT03748771/Prot_SAP_000.pdf